CLINICAL TRIAL: NCT00988832
Title: A UK Retrospective Audit of Patients With Crohn's Disease Treated With Infliximab
Brief Title: An Audit of Patients With Crohn's Disease Treated With Infliximab (P06066)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P06066
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Infliximab: Infliximab as prescribed by a physician in normal practice for Crohn's disease
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab as prescribed by a physician in normal practice for Crohn's disease
  Other Names: Remicade; SCH 215596

SUMMARY:
The aim of this study is to quantify how infliximab therapy is being used in the UK and the consequent impact on health care resources, which will help to inform budget holders and payers on the costs associated with the treatment of Crohn's Disease.

DETAILED DESCRIPTION:
All interested hospital physicians across the UK who prescribe infliximab as part of their treatment of Crohn's Disease patients. will be included. It is assumed that the physician population will consist primarily of gastroenterologists, though general physicians (hospital-based) with an interest in Crohn's Disease may also be included.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's Disease.
* Over the age of 18 years.
* Must have received the first infusion of infliximab on or after 1st January 2003 (when the maintenance therapy license was granted).
* Must have received at least one infusion of infliximab.
* A minimum of 12 months data prior to, and 24 months data post infliximab exposure should be available in the medical records.
* Must have been under the care of the participating center for the entirety of the study period.

Exclusion Criteria:

* Should not have been involved in any clinical trial during the observational period (ie, a minimum of 12 months before and 24 months after first receiving infliximab).
* Should not have received any biologic therapy prior to infliximab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All interested hospital physicians across the UK who prescribe infliximab as part of their treatment of Crohn's Disease patients will be included. Physicians will record information from the medical records of patients who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No subjects were recruited for this retrospective study; participating investigators reviewed medical records of qualifying subjects and provided data to the sponsor.
Groups:
- Infliximab: Infliximab as prescribed by a physician in normal practice for Crohn's disease: 5 mg/kg or 10 mg/kg infusion as either maintenance or episodic therapy.
Period: Overall Study
Arm/Group | Infliximab
Started | 380
Completed | 380
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 380
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at first infusion of infliximab
  years | 37 (13)
Sex/Gender, Customized [Number; unit: participants]
  Female | 208
  Male | 171
  Not Specified | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Cost Per Participant of Consultations With Health Care Providers (HCPs)
Description: Costs were calculated as those incurred to the National Health Service (NHS) to treat Crohn's Disease. Costs of outpatient consultations are based on the 2009 Unit Cost of Health and Social Care published by the Personal Social Service Research Unit. Consultations with gastroenterologists, gastric/gastrointestinal surgeons, radiologists, nurses/Inflammatory Bowel Disease nurses, dieticians/nutrition specialists, psychologists/psychiatrists, pharmacists, and occupational therapists are included in the analysis.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Groups:
- 0-12 Months Pre-Infliximab: Data from the 12 months prior to participants' first infusions of infliximab
- 0-12 Months Post-Infliximab: Data from the first 12 months following participants' first infusions of infliximab
- 0-18 Months Post-Infliximab: Data from the first 18 months following participants' first infusions of infliximab
- 0-24 Months Post-Infliximab: Data from the first 24 months following participants' first infusions of infliximab
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 913.48 (516.36) | 962.30 (547.89) | 1317.58 (730.45) | 1664.45 (910.45)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p < 0.0001, ANOVA

2. Primary Outcome: Mean Cost Per Participant of Elective Surgical Procedures
Description: Costs were calculated as those incurred to the National Health Service (NHS) to treat Crohn's Disease. Costs of elective surgical procedures were calculated as per the 2009 Healthcare Resource Group (HRG) descriptors. Costs were analyzed for elective surgeries that required participants to be admitted into a hospital.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 752.46 (2162.95) | 572.75 (1846.60) | 818.46 (2167.24) | 1078.47 (2484.84)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p = 0.0004, ANOVA

3. Primary Outcome: Mean Cost Per Participant Due to Non-elective/Emergency Inpatient Admissions
Description: Costs were calculated as those incurred to the National Health Service (NHS) to treat Crohn's Disease. Costs of non-elective or emergency inpatient admissions were calculated as per the 2009 Healthcare Resource Group (HRG) descriptors. Costs were analyzed for unplanned hospital admissions due to emergency surgical procedures and unplanned consultations due to complications.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 1107.65 (1979.67) | 769.95 (1831.80) | 1002.33 (2107.25) | 1261.42 (2347.89)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p = 0.0041, ANOVA

4. Primary Outcome: Mean Cost Per Participant for Admissions for Day Case Surgery
Description: Costs were calculated as those incurred to the National Health Service (NHS) to treat Crohn's Disease. Costs of day case (outpatient) surgeries were calculated as per the 2009 Healthcare Resource Group (HRG) descriptors. Costs were analyzed for any surgeries that did not require the participant to stay overnight in the hospital.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 48.73 (247.92) | 18.60 (159.00) | 33.16 (206.28) | 48.13 (260.52)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p = 0.0423, ANOVA

5. Primary Outcome: Mean Cost Per Participant for All Hospitalizations
Description: Costs for all hospitalizations, including costs associated with elective
  and emergency (non-elective) admissions as well as outpatient procedures.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 1908.85 (3092.15) | 1361.30 (2859.93) | 1853.95 (3364.42) | 2388.01 (3885.02)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p = 0.0006, ANOVA

6. Primary Outcome: Mean Cost Per Participant of Accident and Emergency (A&E) Visits
Description: Costs for visits to A&E without admission. Costs were calculated as those incurred to the National Health Service (NHS) to treat Crohn's Disease as per the 2009 Healthcare Resource Group (HRG) descriptors.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 3.01 (18.66) | 4.34 (24.24) | 6.60 (29.57) | 8.22 (35.22)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p = 0.0014, ANOVA

7. Primary Outcome: Mean Cost Per Participant for Crohns-related Medications
Description: Costs of biologics were calculated by multiplying the number of vials of drug used per participant by the 2009 British National Formulary (BNF) cost per vial. Costs of other drugs with ≥10 prescriptions were calculated by multiplying the 2009 BNF daily cost of the standard/most-prescribed dose of the most-prescribed drug (reference drug) in each drug group (Anatomical Therapeutic Classification [ATC] Level 4) by the length of treatment. Costs for drugs in drug groups with ≤9 prescriptions were calculated using the average cost of all Crohns medications multiplied by the length of treatment.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant
  Excluding Biologics | 327.98 (362.36) | 431.78 (485.98) | 653.31 (727.71) | 879.05 (957.98)
  Including adalimumab | 327.98 (362.36) | 615.23 (1163.99) | 1092.65 (2304.38) | 1678.72 (3630.93)
  Including adalimumab and infliximab | 327.98 (362.36) | 9430.57 (4769.30) | 12644.40 (7138.18) | 15934.80 (9616.83)

8. Primary Outcome: Mean Cost Per Participant for Diagnostic Tests During Planned Outpatient Consultations
Description: Costs were calculated as those incurred to the National Health Service (NHS) to treat Crohn's Disease. Costs of diagnostic tests conducted during outpatient consultations were calculated as per the 2008-2009 NHS Reference Costs. Costs for diagnostic tests during hospitalizations and A&E visits were incorporated into cost analyses for those categories and are not included here.
Time Frame: 12 months prior to and 12, 18, and 24 months after the first infusion of infliximab
Measure: Mean (Standard Deviation); unit: Pounds sterling per participant
Arm/Group | 0-12 Months Pre-Infliximab | 0-12 Months Post-Infliximab | 0-18 Months Post-Infliximab | 0-24 Months Post-Infliximab
Number analyzed (Participants) | 380 | 380 | 380 | 380
Pounds sterling per participant | 411 (397.72) | 199.77 (374.94) | 303.94 (480.03) | 380.08 (535.19)
Statistical Analysis 1: Comparison: 0-12 Months Pre-Infliximab vs 0-12 Months Post-Infliximab vs 0-18 Months Post-Infliximab vs 0-24 Months Post-Infliximab; Test type: Superiority or Other; p < 0.0001, ANOVA

ADVERSE EVENTS:
Groups:
- INFLIXIMAB, RECOMBINANT: Infliximab as prescribed by a physician in normal practice for Crohn's disease: 5 mg/kg or 10 mg/kg infusion as either maintenance or episodic therapy.
Arm/Group | INFLIXIMAB, RECOMBINANT
Serious Adverse Events (participants affected / at risk) | 36/380
Other Adverse Events (participants affected / at risk) | 0/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFLIXIMAB, RECOMBINANT (N=380)
HAEMOLYTIC URAEMIC SYNDROME (Blood and lymphatic system disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 2 (2)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1)
FEELING HOT (General disorders) | 1 (1)
MALAISE (General disorders) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 3 (3)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 2 (2)
ANAL ABSCESS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2)
LIVER ABSCESS (Infections and infestations) | 1 (1)
MENINGITIS HERPES (Infections and infestations) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
TRACHEOBRONCHITIS (Infections and infestations) | 1 (2)
DRUG EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 3 (3)
DRUG EXPOSURE VIA BREAST MILK (Injury, poisoning and procedural complications) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 8 (8)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
ANTINUCLEAR ANTIBODY POSITIVE (Investigations) | 1 (1)
HEART RATE INCREASED (Investigations) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
MYELITIS TRANSVERSE (Nervous system disorders) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CUTANEOUS LUPUS ERYTHEMATOSUS (Skin and subcutaneous tissue disorders) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognises the right of the investigator to publish the study results. The investigator is asked to send a draft of the publication/abstract to the Sponsor 30 days in advance of submission in order to obtain approval prior to submission. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion, the contents of the publication will be discussed in order to find a solution which satisfies both parties.